CLINICAL TRIAL: NCT00117520
Title: The Effect of Caffeine as Endurance Enhancing Drug in the Elderly
Brief Title: The Effect of Caffeine in Elderly Citizens
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Herning Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2612-1987
Record Dates: First submitted 2005-06-30; First posted 2005-07-07 (Estimated); Last update posted 2006-07-07 (Estimated); Status verified 2002-07

CONDITIONS: Healthy Elderly Citizens
Keywords: caffeine, endurance, postural stability, elderly
MeSH Terms: interventions — Caffeine

INTERVENTIONS:
Drug: Caffeine

SUMMARY:
The study investigated the effect of caffeine on physical performance in healthy citizens aged over 70 years. The main hypothesis was that 6 mg/kg caffeine would improve cycling endurance at 65% of expected maximal heart rate.

DETAILED DESCRIPTION:
Caffeine ingestion increases the endurance of young people exercising at 60%-85% of their maximal oxygen uptake, and it also seems to improve endurance as measured by repeated sub-maximal isometric contraction and decreases the rate of perceived exertion during exercise. Although caffeine increases endurance in young people, an increase in endurance may be of greater interest in the elderly as the population of older adults with a physically active lifestyle is growing rapidly or for increasing endurance fitness through an exercise or rehabilitation program. Therefore the main hypothesis was that caffeine would improve cycling endurance at 65% of expected maximal heart rate, and the secondary hypotheses were that caffeine would improve postural stability, reaction and movement times, isometric arm flexion endurance, and walking speed, and would reduce the rate of perceived exertion after 5 minutes of cycling in healthy elderly citizens.

ELIGIBILITY:
Inclusion Criteria:

* Healthy elderly individuals aged over 70 years

Exclusion Criteria:

* Dementia or invalidating psychiatric disease
* General debility, angina, or other diseases that would render participation in the test program impossible
* Treatment with beta receptor blocking drugs, calcium-channel blocking drugs, digitalis, or nitroglycerine
* Acute disease and injury
* Diabetes
* Conditions that would contraindicate caffeine ingestion or participation in the test program
* Treatment with medication that interacts with caffeine
* Ingestion of caffeine containing drinks and foods 48 hours before each session

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30
Dates: Start 2002-07; Study Completion 2006-03

PRIMARY OUTCOMES:
endurance measured on an ergometer bicycle

SECONDARY OUTCOMES:
postural stability
reactiontime
isometric endurance (armflexion)
walking speed
fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte B Norager, M.D, Principal Investigator — Surgical Research Department, Herning Hospital, DK-7400 Herning
Locations (1):
- Surgical Research Department, Herning, Ringkjoebing, Denmark